CLINICAL TRIAL: NCT03947567
Title: A Multicenter, Open, Extension Trial to Evaluate Safety and Efficacy of Recombinant Human Coagulation Factor VIII (SCT800) During Long Term Treatment in Previously Treated Patients With Severe Haemophilia A .
Brief Title: Safety and Efficacy of Long-term Treatment With SCT800 in Previously Treated Hemophilia A Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SCT800-A401
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant Human Coagulation FVIII (Experimental)
  Interventions: Drug: Recombinant Human Coagulation FVIII

INTERVENTIONS:
Drug: Recombinant Human Coagulation FVIII — Participants received SCT800 for prophylaxis and/or on-demand treatment for 120 weeks.
  Other Names: SCT800

SUMMARY:
This study is a multi-center, open-label, extension trial to evaluate the safety, efficacy of SCT800 in long term prophylaxis and on-demand treatment in patients with severe hemophilia A who have been previously treated with coagulation factor VIII(FVIII) . This study includes two phases: the screening period and prophylaxis period.Prophylaxis with 25 - 50 IU/kg of SCT800 shall be administered once every other day or three times per week starting from V1, on-demand treatment is given when bleeding episodes occur. The study period is 120 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male patients who are diagnosed with severe (laboratory tested FVIII:C <2%) hemophilia A;
* Patients Who Completed trial of SCT800-A302 or SCT800-A 303 and New PTP(previously treated patients)(Previously received FVIII prophylactic or bleeding treatment, have the relevant records and are verified to have accumulated exposures days( EDs) ≥150 days;
* Negative FVIII inhibitor assay results (laboratory tested Nijmegen-Bethesda assay result <0.6 BU(Bethesda unit)/mL);
* The treatment records of at least 50EDs before screening can be obtained;
* HIV negative; if HIV positive, the viral load <200 particles/uL or <400,000 copies/mL, and HIV patients must satisfy CD4+ count >200/μL;
* The patient or his guardian voluntarily signed the Informed Consent Form.

Exclusion Criteria:

* Known allergy to any coagulation factor VIII or any excipient; known allergy to bovine, rodent or hamster bovine;
* Has a history or family history of blood coagulation factor VIII inhibitor;
* Patients with other coagulation dysfunction diseases in addition to hemophilia A;
* Patients with other clinically significant diseases, alcoholism, drug abuse, mental disorders or intellectual disabilities;
* Patients with other severe or clinical significant diseases verified by the investigator to be unable to benefit from the clinical study;
* Patients who participated in other clinical studies within one month before the first drug administration (except FVIII trials) and patients who participated in other FVIII clinical trials after signing the Informed Consent Form;

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Hemophilia A is a kind of sex chromosome recessive genetic disease and ofter occurs in male.
Enrollment: 240 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of FVIII inhibitors | up to 120 weeks
  The Nijmegen-Bethesda assay shall be used to monitor the production of FVIII inhibitors during the trial.

SECONDARY OUTCOMES:
Annualized Bleeding Rate | up to 120 weeks
  Annualized Bleeding Rate（ABR） can be calculated using the following formula: Number of bleeding events in efficacy evaluation period/(number of days in treatment period/365.25)
FVIII incremental in-vivo recovery | up to 120 weeks
  Incremental recovery is determined as the peak factor level recorded in the first hour after infusion and is reported as [IU/ml]/[IU/kg]
Bleeding event treatment efficacy | up to 120 weeks
  The investigator shall evaluate the hemostatic effect after the treatment of every bleeding event of subjects based on a four-point scale(excellent, good, moderate, not relieved).

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China